CLINICAL TRIAL: NCT01387308
Title: An Open-label, Partially Randomized, 5-way Crossover Study in Healthy Volunteers to Assess the Relative Bioavailability of 100 and 150 mg Fostamatinib Tablets Compared With 50 mg Fostamatinib Tablets
Brief Title: Study in Healthy Males to Assess the Bioavailability of 4 Different Fostamatinib Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00018
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Phase 1; Healthy male volunteers; pharmacokinetics; fostamatinib; Scientific Terminology: Bioavailability, R406 plasma AUC and C_maxR406 plasma AUC0-t, t1/2λz and t_max; Laymen Terminology: Amount of R406 in blood
MeSH Terms: interventions — fostamatinib

ARMS (5):
- A (Experimental): Fostamatinib 50 mg tablet x 2 (Phase 3 batch)
  Interventions: Drug: Fostamatinib
- B (Sham Comparator): Fostamatinib 50 mg tablet x 3 (Phase 3 batch)
  Interventions: Drug: Fostamatinib
- C (Experimental): Fostamatinib 100 mg tablet (new formulation)
  Interventions: Drug: Fostamatinib
- D (Experimental): Fostamatinib 150 mg tablet (new formulation)
  Interventions: Drug: Fostamatinib
- E (Experimental): Fostamatinib 50 mg tablet x 2 (Phase 3 batch)
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Oral tablets, 50 mg x 2, single dose
  Arms: A
Drug: Fostamatinib — Oral tablets, 50 mg x 3, single dose
  Arms: B
Drug: Fostamatinib — Oral tablets, 100 mg, single dose
  Arms: C
Drug: Fostamatinib — Oral tablets, 150 mg, single dose
  Arms: D
Drug: Fostamatinib — Oral tablets, 50 mg x 2, single dose
  Arms: E

SUMMARY:
Study in healthy males to assess bioavailability of 4 different fostamatinib tablets.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent prior to any study specific procedures
* Volunteers will be males aged 18 to 55 years and with a weight of at least 50 kg and body mass index (BMI) between 18 and 30 kg/m2 inclusive
* Volunteers agreeing to participate in the optional genetic research must provide a separate, signed, written and dated informed consent for genetic research. The volunteer will not be excluded from other aspects of the study described in this Clinical Study Protocol so long as they consent to them

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product
* Subjects who smoke more than 5 cigarettes or the equivalent in tobacco per day
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess the relative bioavailability of R406 in healthy volunteers when fostamatinib is administered as a reformulated 100-mg tablet versus 2 x 50-mg tablets (Phase III formulation) | From Pre-dose until 96 hours post dose of each treatment period
  Assessments will include but is not limited to: plasma R406 AUC, Cmax
To assess the relative bioavailability of R406 in healthy volunteers when fostamatinib is administered as a reformulated 150-mg tablet versus 3 x 50-mg tablets (Phase III formulation) | From pre-dose until 96 hours post dose of each treatment period
  Assessments will include but is not limited to: plasma R406 AUC, Cmax )

SECONDARY OUTCOMES:
To examine the safety and tolerability of fostamatinib 50 mg, 100 mg, and 150 mg tablet batches | From pre-dose until 96 hours post dose of each treatment period
  The safety endpoints will include adverse event monitoring, vital signs, physical examinations, clinical laboratory tests, ECGs.
To estimate the within subject variability in R406 exposure when fostamatinib 50 mg tablets are administered on 2 separate occasions. | From pre-dose until 96 hours post dose of each treatment period
  Assessments will include but is not limited to: plasma R406 plasma AUC0-t, t1/2, and tmax

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States